CLINICAL TRIAL: NCT05190094
Title: Multicenter, First-line Metastatic Open-label Prospective Phase II Trial Evaluating the Combination of Palbociclib (CDK 4/6 Inhibitor) and Hormone Therapy (Letrozole or Anastrozole) in Women With Luminal, HER2 Negative Advanced Breast Cancer: Evaluation of the Prediction of Individual Treatment Efficacy Using Infrared Laser Spectroscopy Analysis on Liquid Biopsies (Quantum Optics).
Brief Title: Prediction of Treatment Efficacy of the Combination of Palbociclib/(Letrozole or Anastrozole) in First Line Metastatic Women With Luminal, HER2 Negative Advanced Breast Cancer, Using Infrared Laser Spectroscopy Analysis on Liquid Biopsies.
Acronym: ICRG0201
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Cancer Research Group, United Arab Emirates (Other)
Collaborators: King Saud Medical City (Other Government); Max-Planck-Institut für Quantenoptik (MPQ), and Faculty of Physics at Ludwig-Maximilians-Universität München (LMU), Garching, Germany (Unknown); King Abdallah University for Science and Technology (KAUST), Thuwal, Saudi Arabia. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICRG0201
Record Dates: First submitted 2021-12-08; First posted 2022-01-13 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-03

CONDITIONS: Hormonal Receptors Positive, HER2 Negative, Advanced Breast Cancer
MeSH Terms: interventions — Aromatase Inhibitors; Letrozole; Anastrozole

STUDY DESIGN:
Intervention Model Description: This is a multicenter, open-label study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Palbociclib + Aromatase Inhibitors (AI) (Letrozole or Anatrozole) (Experimental): The participants will receive a combination of: Palbociclib (125 mg daily per os (3 weeks on-1 week off) with dose adaptation according to safety profile) and non-steroidal aromatase inhibitor (Letrozole (2.5mg ) or Anastrozole (1mg) daily per os). This combination will continue until progression for an average duration of 2 years.
  Interventions: Drug: Combination of Palbociclib and aromatase inhibitor (Letrozole or Anastrozole)

INTERVENTIONS:
Drug: Combination of Palbociclib and aromatase inhibitor (Letrozole or Anastrozole) — A combination of Palbociclib (125 mg daily per os (3 weeks on-1 week off) with dose adaptation according to safety profile) and non-steroidal aromatase inhibitor (Letrozole (2.5mg ) or Anastrozole (1mg) daily per os).

SUMMARY:
This study is a multicenter, international, open-label phase II study. Based on inclusion/exclusion criteria, eligible pre and postmenopausal patients with newly diagnosed metastatic luminal hormone receptor-positive and HER2 negative breast cancer, will be prospectively treated with a standard combination of hormone therapy (Letrozole or Anastrozole) and Palbociclib. This combination will continue until progression. Treatment response will be evaluated every three months using clinical and radiological assessments (Revised RECIST guidelines).

Patients will undergo serial liquid biopsies (blood tests) for plasma molecular fingerprinting by the Quantum Optics technology. This study will be the first program exploring the adjunction of the Quantum Optics technology on liquid biopsies to define individual 'molecular fingerprinting profiles' to predict the individual therapeutic effects of Palbociclib combined with Aromatase Inhibitors (AI) (plus ovarian function suppression (OFS) for pre/peri-menopausal patients) in luminal hormone receptor-positive and HER2 negative advanced breast cancer. Batteries of algorithmic tests will integrate the variables obtained by Quantum Optics (to evaluate the efficacy or not of the combination of Palbociclib + Aromatase Inhibitors (AI) ). This approach introduces the concept of singularity to break from the classic idea of "one size fits all".

DETAILED DESCRIPTION:
Background:

The standard therapy of first-line metastatic luminal hormone receptor positive, HER2 negative breast cancer, is based upon the combination of hormone therapy (HT): an aromatase inhibitor (AI) (e.g. Anastrozole or Letrozole) and a CDK 4/6 inhibitor (e.g. Palbociclib). Around 50% of patients are benefiting from this combination. However, there are no predictive markers to identify upfront the benefiting population, thus imposing to treat the whole population (100%) for the benefit of 50%.

Objectives:

Primary:

* Rate of objective clinical response for the combination of Palbociclib + AI.
* Value of quantum optics (QO) analysis on liquid biopsies to predict the upfront efficacy/resistance of the combination (Palbociclib + AI) on an individual basis.

Secondary:

* Progression-Free Survival (PFS).
* Clinical benefit (CR/PR/Stabilization>24 weeks).
* 'Objective' clinical benefit (CR/PR/Minor response (> 0% > 24 weeks).
* Modification of the individual molecular fingerprinting during treatment.
* Role of individualized molecular fingerprinting to predict early progression (>6 months).
* Role of individualized molecular fingerprinting to predict relapse in age-matched patients with an initial response.
* Safety and tolerability of the proposed regimen.
* Benchmark analysis, using Raman Spectroscopy.

Materials and Methods:

Study design:

This study is a multicenter, international, open-label phase II study. Based on inclusion/exclusion criteria, eligible pre and post-menopausal patients with newly diagnosed metastatic Luminal HER2 negative breast cancer, will be prospectively treated with a standard combination of HT (AI: Letrozole or Anastrozole) and Palbociclib. This combination will continue until progression. Treatment response will be evaluated every three months using clinical and radiological assessments (Revised RECIST guidelines).

Patients will undergo liquid biopsies (blood tests) for plasma molecular fingerprinting by the QO technology at enrolment, each month for the first three months and then every three months until relapse, along with clinical and radiological assessments every three months.

Sample size: Considering the approximately 50% response rate (RR) previously reported in the phase III PALOMA 2 trial (AI + Palbociclib) and the initial published data of QO analysis on liquid biopsies, which compared plasma molecular fingerprint profiles between a control population without breast cancer and a population with breast cancer (sensitivity: 98% / specificity: 97%), we hypothesize that the sensitivity to differentiate responders to non-responders by QO analysis on liquid biopsies (prediction of efficacy) will be 97%. Based on the above hypothesis, the sample size calculated using alpha 5% and power 95% is N=80 patients to be enrolled and treated.

Populations:

The Intent-to-Treat (ITT): all patients enrolled in the study. The safety population: all patients receiving any treatment.

Statistical Methodology:

Qualitative variables are frequency and percentage. Comparison of the proportion between responders and non-responders will use the chi-square test.

Quantitative variables: mean, standard deviation, median, maximum, and minimum. Time-dependent parameters: Kaplan-Meier method. Cox's proportional hazards regression analysis for response rates, clinical benefits, PFS.

All tests of hypotheses: one-sided. Confidence intervals of the median survival: method of Simon.

The methodology of computational analysis: "non-hierarchical deep data mining" approach with:

* Analyses with the support vector machines with a polynomial nucleus.
* Age stratifications when applicable with sub-stratifications in different age groups.

ELIGIBILITY:
Inclusion Criteria:

To be enrolled in the study, patients should meet the following inclusion criteria:

1. Written informed consent before beginning specific protocol procedures including expected cooperation of the patients for the treatment and follow-up must be obtained and documented according to the local regulatory requirements.
2. Postmenopausal women or pre/peri-menopausal women with Surgical oophorectomy (preferred) or Analogs of LHRH.
3. Performance status < 3 (according to WHO criteria).
4. Histologically confirmed breast cancer (Luminal A or B).
5. Estrogen Receptor positive (ER > 1%).
6. HER2 negative (score 0 or 1 by immunochemistry), FISH negative if IHC score 2.
7. Clinical stage IIIb & IV.
8. Either:

   1. Women with De novo advanced luminal HER2 negative advanced breast cancer without other prior systemic treatment for advanced disease.
   2. Women with luminal HER2 negative advanced breast cancer either with secondary resistance (relapse after 2 years of adjuvant hormone therapy or within 12 months of completion of adjuvant HT) or sensitivity to adjuvant HT (relapse > 12 months after completion of adjuvant HT).
9. Measurable or evaluable disease.
10. Hematology:

    * Neutrophil count ≥ 1.5 G/L,
    * Platelet count ≥ 100 G/L,
    * Leucocyte count > 3.0 G/L,
    * Hb> 9g/dl.
11. Hepatic function:

    * Total bilirubin ≤ 1.5 times the upper normal limit (UNL),
    * ASAT ≤ 2.5xUNL,
    * ALAT ≤ 2.5xUNL,
    * Alkaline phosphatase ≤ 2.5 times the upper normal limit (UNL).
12. Renal function:

    • Serum creatinine ≤1.5xUNL (and if Serum creatinine >1.5xUNL, creatinine clearance ≥40 mL/min),
13. Metabolic function:

    • Serum calcium ≥ lower limit of normal.
14. Negative pregnancy test (urine or serum) within 7 days before registration for all women of childbearing potential. Patients of childbearing potential must implement adequate non-hormonal contraceptive measures during study treatment.
15. Patients with negative Human Immunodeficiency Virus (HIV) and/or Hepatitis B and/or Hepatitis C results.

Exclusion Criteria:

To be enrolled in the study, patients should meet the following exclusion criteria:

1. Male patients.
2. HER2 positive tumors or unknown HR/HER2 status.
3. Triple-negative Breast Cancer (ER<1%).
4. Pregnant or breast-feeding women, or those who plan to become pregnant within 6 months post-treatment.
5. No willingness to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months post-treatment.
6. Any form of breast cancer other than those described in the inclusion criteria, particularly inflammatory and/or loco-regional disease (stages I, II & IIIa).
7. Non-evaluable tumor.
8. Bilateral breast cancer.
9. Patients with a history of other cancer, except in situ cervical cancer or baso-cellular skin cancer, considered cured.
10. Patient has another disease, which is deemed incompatible with the inclusion in the protocol.
11. Heart, kidney, medullary, respiratory or liver failure.

    * Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) at baseline.
    * History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease at baseline,
    * Acute urinary infection, ongoing hemorrhagic cystitis at baseline.
12. Uncontrolled diabetes.
13. Symptomatic or progressive disorder of the central nervous system (CNS) at baseline.
14. Patients with positive Human Immunodeficiency Virus (HIV) and/or Hepatitis B and/or Hepatitis C results.
15. Significant psychiatric abnormalities.
16. History of hypersensitivity to studied treatment or excipients.
17. Known previous or ongoing abuse of narcotic drug, other medication or alcohol.
18. Any investigational agent within 30 days before initiation of study treatment.
19. Patient unwilling or unable to comply with study requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-12-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of Objective Clinical Response | From date of first treatment until the date of the first documented progression, assessed up to 2 years.
  The objective clinical response will be assessed with Radiological evaluation according to the RECIST revised criteria for the combination of Palbociclib + Aromatase Inhibitors (AI)
Sensitivity and Specificity of prediction of the efficacy of the combination (palbociclib +AI). | From date of first treatment until the date of the first documented progression, assessed up to 2 years.
  Sensitivity and specificity of infrared laser spectroscopy analysis on liquid biopsies to predict the efficacy/resistance of the combination (Palbociclib + Aromatase Inhibitors (AI)) on an individual basis.

SECONDARY OUTCOMES:
Rate of Progression-Free Survival (PFS) | From Baseline to time of progression for an average duration of 2 years.
  Progression-Free Survival (PFS)
Rate of Clinical benefit | From time CR/PR/Stabilization up to more than 24 weeks
  Clinical benefit is defined as CR/PR/Stabilization for more than 24 weeks
Rate of 'Objective' clinical benefit | From time CR/PR/Minor response [> 0%] up to more than 24 weeks
  'Objective' clinical benefit is defined as CR/PR/Minor response [> 0%] more than 24 weeks).
Modification of the individual molecular fingerprinting | From the date of first treatment until the date of the first documented progression, assessed up to 2 years.
  Modification of the individual molecular fingerprinting
Prediction of progression in patients with initial response and objective clinical benefit | From the date of first treatment until the date of the first documented progression, assessed up to 2 years.
  Modification of individualized molecular fingerprinting will be used to predict progression
Prediction of progression in age-matched patients with initial response and objective clinical benefit | From the date of first treatment until the date of the first documented progression, assessed up to 2 years.
  Modification of individualized molecular fingerprinting will be used to predict progression
Prediction of early progression (>6 months). | During the course of study treatment, after M6 up to an average duration of 2 years.
  Modification of individualized molecular fingerprinting will be used to predict early progression (>6 months).
Number of patients with related adverse reactions | During the course of study treatment until progression, for an average duration of 2 years.
  Adverse events will be collected during the course of the study. Relationship to study drug is also reported.
Prediction of Progression obtained from Raman spectroscopy | From the date of first treatment until the date of the first documented progression, assessed up to 2 years.
  Modification of individualized molecular fingerprinting will be used to predict progression obtained from Raman spectroscopy as a benchmark analysis

CONTACTS AND LOCATIONS:
Overall Officials: M.R.K. BAHADOOR, MD, EMBA, Study Director — International Cancer Research Group
Locations (7):
- Algeria (2):
  - EHS LCC Blida, Medical Oncology Center, Blida
  - University Hospital Sétif,, Sétif
- King Hussein Cancer Center (KHCC) - Amman, Amman, Jordan
- Saudi Arabia (4):
  - King Saud Medical City - KSMC, Riyadh
  - Medical Oncology Center- King Saud University Medical City (KSUMC), Riyadh
  - Medical Oncology Department- King Fahad Medical City (KFMC), Riyadh
  - Oncology Center Department, King Faisal Specialist Hospital and Research Centre -KFSH & RC, Riyadh

IPD SHARING:
Plan to Share IPD: No